CLINICAL TRIAL: NCT01312220
Title: Relationship of Serological Growth Factors and Hepatic Progenitor Cells in Acute Liver Failure
Brief Title: Growth Factors and Hepatic Progenitor Cells in Acute Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: CM Ho, NTUH
Other Study IDs: 201101061RC
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-02

CONDITIONS: the Focus of the Study is to Correlate the Growth Factors in Serum With the Progenitor Cells in Liver

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Serum Liver piece

SUMMARY:
To study the correlation of serological growth factors and the hepatic progenitor cells involved in liver regeneration of liver failure.

ELIGIBILITY:
Inclusion Criteria:

Acute liver failure Received iver transplantation

Exclusion Criteria:

Pregnancy Sepsis Heart failure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute liver failure who received liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-02; Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: CM Ho, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan, Taiwan